CLINICAL TRIAL: NCT06506656
Title: Effect of an Intra-articular Treatment With a Combination of Hyaluronic Acid and Adelmidrol (Hyadrol®) on Pain, Joint Stiffness and Functional Limitation in Patients With Degenerative Joint Disease
Brief Title: Hyaluronic Acid and Adelmidrol (Hyadrol®) in Patients With Degenerative Joint Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Azienda Ospedaliera "Sant'Andrea" (Other)
Responsible Party: Principal Investigator, Maria Chiara Vulpiani, Associate Professor, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hy-ad2
Record Dates: First submitted 2024-07-01; First posted 2024-07-17 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Degenerative Joint Disease
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with coxarthrosis (Experimental): Three intra-articular infiltrations (1/week) with 2 ml Hyaluronic Acid and Adelmidrol
  Interventions: Device: Hyadrol®
- Patients with rhizoarthrosis (Experimental): Three intra-articular infiltrations (1/week) with 1 ml Hyaluronic Acid and Adelmidrol
  Interventions: Device: Hyadrol®

INTERVENTIONS:
Device: Hyadrol® — Sterile single-use Medical Device for intra-articular injections

SUMMARY:
Osteoarthritis is a major cause of chronic musculoskeletal pain. Behind this disorder there is a process of chronic neuroinflammation due to the overactivation of mast cells at the tissue level. The mast cells present in the synovial membranes act as first sensors in pathological situations, degranulating in an uncontrolled manner.

Furthermore, in degenerative joint pathologies, there is a marked reduction in the viscoelastic capacity of the synovial fluid associated with a reduction in both the concentration and the average molecular weight of endogenous hyaluronic acid. The association of hyaluronic acid and Adelmidrol (Hyadrol®) could represent an effective treatment for controlling the neuroinflammation process that supports degenerative joint diseases.

The objective of the present clinical investigation is to evaluate its safety and efficacy in patients with arthritis of the hip (coxarthrosis) and trapezium-metacarpal joints (rhizoarthrosis).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 40 years;
* both genders;
* diagnosis of stage II-III coxarthrosis or rhizoarthrosis according to radiological classification (Kellgren and Lawrence or modified Eaton-Littler criteria respectively)
* pain intensity ≥ 5 on NRS;
* wash-out for at least two weeks from anti-inflammatory drugs before enrollment;
* compliant patients;
* signed informed consent.

Exclusion Criteria:

* age < 40 years;
* presence of concomitant inflammatory systemic pathologies (e.g.: rheumatoid arthritis, etc.);
* severe and progressive clinical conditions,
* NSAIDs therapy in the 2 weeks prior to enrollment;
* corticosteroid therapy in the 3 months prior to enrollment;
* chondroprotectors intake in the 6 months prior to enrollment;
* arthroscopic procedures or intra-articular visco-supplementation in the 6 months prior to enrollment;
* presence of cognitive impairment;
* ongoing rehabilitation and/or physiotherapy;
* allergy or hypersensitivity to the study treatment;
* pregnant and/or lactating female subjects;
* not compliant patients;
* denied informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change of degenerative joint disease symptoms in patients with coxarthrosis: | Baseline (T0): first intra-articular infiltration; Treatment (T1): second intra-articular infiltration; Treatment (T2): third intra-articular infiltration; Follow up (T3): 1 week after T2; Follow up (T4): 4 weeks after T3
  Evaluation of degenerative joint disease symptoms assessed by Western Ontario and McMaster Universities (WOMAC) scale for patients with coxarthrosis. WOMAC is a self-report questionnaire consisting of 24 questions divided into 3 groups: pain (5 items), joint stiffness (2 items) and functional limitations (17 items). Each question has 5 possible answers, evaluate in a Likert scale, from 0 (none) to 4 (extreme):
  * pain: score from 0 to 20;
  * joint stiffness: score from 0 to 8;
  * functional limitations: score from 0 to 68.
  The sum of the individual scores results in an overall score from 0 to 96 (96 indicates severe disability).
Change of degenerative joint disease symptoms in patients with rhizoarthrosis: | Baseline (T0): first intra-articular infiltration; Treatment (T1): second intra-articular infiltration; Treatment (T2): third intra-articular infiltration; Follow up (T3): 1 week after T2; Follow up (T4): 4 weeks after T3
  Evaluation of degenerative joint disease symptoms assessed by Disabilities of the Arm, Shoulder and Hand (DASH) questionnaires for patients with rhizoarthrosis.The questionnaire is divided into 3 modules: symptom/disability module consisting of 30 questions investigating aspects of daily life; occupational module and sports/recreational activities module (optional) consisting of 8 questions in total. Optional items are used for workers and individuals whose occupation or sports or recreational activity requires a high level of physical performance. Each question has 5 possible answers, from 1 (no difficulty) to 5 (unable to perform a specific activity). The sum of the individual scores results in an overall score, which is converted into a scale from 0 to 100 (100 indicates severe disability).

SECONDARY OUTCOMES:
Change of pain symptoms: | Baseline (T0): first intra-articular infiltration; Treatment (T1): second intra-articular infiltration; Treatment (T2): third intra-articular infiltration; Follow up (T3): 1 week after T2; Follow up (T4): 4 weeks after T3
  Evaluation of pain intensity assessed by the 11-point Numeric Rating Scale (NRS) scored from 0 to 10, where 0 indicates 'no pain' and 10 corresponds to 'the worst pain ever possible'. The higher the score, the more severe the pain.
Change of patients quality of life: | Follow up (T3): one week after the last infiltration; Follow up (T4): four weeks after T3
  Quality of Life evaluated by the 12-Item Short Form Health Survey (SF-12). The SF-12 is a self-reported health questionnaire. The score produces two summary measures: a mental (MCS-12) and a physical component score (PCS-12). The PCS-12 score is derived from the subdimensions of general health, physical functioning, role physical, and bodily pain, while the MCS-12 score is derived from the subdimensions of social functioning, role emotional, mental health, and energy. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Change of patients self-assessed health status: | Follow up (T3): one week after the last infiltration; Follow up (T4): four weeks after T3
  The patient's global health status is evaluated through the Likert Patient Global Impression of Change (PGIC) scored in 7 points (from 1, very much improved to 7, very much worse).
Incidence of Adverse Events (Safety and Tolerability): | Baseline (T0): first intra-articular infiltration; Treatment (T1): second intra-articular infiltration; Treatment (T2): third intra-articular infiltration; Follow up (T3): 1 week after T2; Follow up (T4): 4 weeks after T3
  Safety of treatment evaluated by monitoring the incidence and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Chiara Vulpiani, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Azienda Ospedaliero-Universitaria Sant'Andrea, Roma, Italy

REFERENCES:
- See also: Guida F et al.,Targeting Neuroinflammation in Osteoarthritis with Intra-Articular Adelmidrol. Biomolecules. 2022; 11;12(10):1453 — https://pubmed.ncbi.nlm.nih.gov/36291664/
- See also: Vulpiani MC et al.,Hyaluronic acid alone versus hyaluronic acid associated with adelmidrol for Intra-articular treatment of knee osteoarthritis: A long-term follow -up. Int J Physiother Res 2023;11(1):4453-4460. — https://www.ijmhr.org/IntJPhysiotherRes/IJPR.2022.192
- See also: Cavallaro C et al.,Adelmidrol Protects Hyaluronic Acid against Oxidative Degradation and Improves the Outcome in Patients with Adhesive Capsulitis of the Shoulder Managed by Physical Therapy. J Orthop Res Ther 2024 — https://www.gavinpublishers.com/article/view/adelmidrol-protects-hyaluronic-acid-against-oxidative--degradation-and-improves-the-outcome-in-patients-with--adhesive-capsulitis-of-the-shoulder-managed-by-physical-therapy-in-vitro-evidence-and-two-case-reports